CLINICAL TRIAL: NCT06629610
Title: A Community-led Intervention (DAiLY) Promoting a Heart-healthy Diet and Active Lifestyle: The Yup'ik Way
Brief Title: Diet and Active Lifestyle - Yuuyaraq (The Yup'ik Way of Life)
Acronym: DAiLY
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: Johns Hopkins Bloomberg School of Public Health (Other); University of Alabama at Birmingham (Other); Marshfield Clinic Research Foundation (Other); University of Alaska Fairbanks (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Bert Boyer, Professor, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01HL168854 (NIH); 1R01HL168854 (NIH)
Record Dates: First submitted 2024-09-30; First posted 2024-10-08 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2024-10

CONDITIONS: Heart Disease
Keywords: Intervention; Alaska Native; Heart Disease; Community Health
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Immediate Intervention (Experimental): This arm is made up of two communities that will receive the intervention at the beginning of the trial. The intervention includes three components, all supported by social media.
  Home-Based Workshops will be delivered by community members to increase knowledge and skills related to food choices, and to emphasize the importance of physical activity. Emphasis is placed on the benefits of consuming subsistence foods, as well as healthy store-bought foods. Food store modifications will increase access to healthy foods in local stores by working with store managers to stock and promote affordable healthy foods, and will provide participants with opportunities to implement what they have learned in workshops. Point of purchase promotions, educational displays, taste tests and cooking demonstrations, will identify and promote these foods. Physical activity promotion will include community-wide traditional activities, such as traditional dance, sports events, and berry festivals.
  Interventions: Behavioral: DAiLY
- Delayed Intervention (Experimental): This arm is made up of two communities that will receive the intervention at the after the immediate arm. The intervention includes three components, all supported by social media.
  Home-Based Workshops will be delivered by community members to increase knowledge and skills related to food choices, and to emphasize the importance of physical activity. Emphasis is placed on the benefits of consuming subsistence foods, as well as healthy store-bought foods. Food store modifications will increase access to healthy foods in local stores by working with store managers to stock and promote affordable healthy foods, and will provide participants with opportunities to implement what they have learned in workshops. Point of purchase promotions, educational displays, taste tests and cooking demonstrations, will identify and promote these foods. Physical activity promotion will include community-wide traditional activities, such as traditional dance, sports events, and berry festivals.
  Interventions: Behavioral: DAiLY

INTERVENTIONS:
Behavioral: DAiLY — The 2-year intervention includes three components, all supported by social media. Home-Based Workshops will be delivered by community members to increase knowledge and skills related to food choices, and to emphasize the importance of physical activity. Emphasis is placed on the benefits of consuming subsistence foods, as well as healthy store-bought foods. Food store modifications will increase access to healthy foods in local stores by working with store managers to stock and promote affordable healthy foods, and will provide participants with opportunities to implement what they have learned in HBWs. Point of purchase promotions, educational displays, taste tests and cooking demonstrations, will identify and promote these foods to community members. Physical activity promotion will include community-wide traditional activities, such as traditional dance, sports events, and berry festivals. Fitbits will be used as a motivational tool for participants to track their progress.

SUMMARY:
Heart disease is the leading cause of death for Alaska Native men and the second leading cause of death (after cancer) among women and Alaska Native people overall. The overarching goal of the proposed multilevel, multicomponent intervention, Diet and Active Lifestyle - Yuuyaraq (DAiLY), is to reduce consumption of highly processed store-bought foods while promoting intake of subsistence foods, healthy store-bought foods, and a more active lifestyle to reduce heart disease risk. The Yup'ik word Yuuyaraq means 'the Yup'ik way of life' and encompasses a worldview in which living in harmony with the environment, as well as sharing of subsistence foods and traditional knowledge is central. The proposed DAiLY intervention is grounded in the Yup'ik worldview and Indigenous Food Sovereignty, and supported by a foundation of trust resulting from 22 years of continuous Community Based Participatory Research on heart disease risk andprotective factors with Yup'ik communities. DAiLY is a direct response to the intervention research requests of community partners and input from Yup'ik Community Research Associates and a Yup'ik Community Planning Group during the formative research and community engagement process shaping this proposal. The proposed intervention, based on the Warnecke model of health disparities and social cognitive theory, includes three components: 1) home-based workshops, framed in the Yupik worldview, led by Community Research Associates to facilitate interactive discussions with community members about healthy market foods, as well as the health benefits of locally harvested traditional foods and increased physical activity; 2) local food store interventions to increase access to, and help build demand for, healthy food options; and 3) traditional community activities, including Yuraq (Yup'ik traditional dance), Native sports events, and berry festivals, that provide opportunities to increase physical activity. The three components will be supported and reinforced via community media, including Facebook, text messaging and visual materials. A continuous metabolic syndrome score will be used as the primary outcome to assess changes in heart disease risk, and objective stable isotope biomarkers of diet and a validated food frequency questionnaire will be used to measure intake of traditional and market foods. We will test the DAiLY intervention in four Yupik communities, randomized to immediate and delayed intervention. Aim 1, will determine the effectiveness of the DAiLY intervention on heart disease risk by measuring change in a continuous metabolic syndrome risk score (primary outcome). Aim 2, will assess implementation of the DAiLY intervention using a mixed methods process evaluation to determine fidelity, dose, and reach, as well as barriers and facilitators to implementation of program activities and participant satisfaction and engagement. Aim 3, will determine the impact of the DAiLY intervention on community-level outcomes, including access to, and sales of, healthy foods in local stores, as well as opportunities for physical activity at community venues.

DETAILED DESCRIPTION:
Background Heart disease (HD) is the leading cause of death for Alaska Native men and the second leading cause of death among women. HD mortality among the Yup'ik Alaska Native people is 30% higher than that for all races in the U.S. The traditional Yup'ik diet is associated with a reduction in multiple risk factors for HD, but over the past 60 years, this dietary pattern has been replaced by a shift toward ultra-processed foods high in saturated fat, salt and sugar which have been linked to increased risk for HD. At the same time, there has been a shift to a more sedentary lifestyle. The goal of this project is to determine the effectiveness of a culturally adapted intervention to reduce HD risk among Yup'ik Alaska Native people by encouraging increased consumption of heart healthy traditional and market foods, as well as increased physical activity.

Intervention Approach This work adheres to a Community-Based Participatory Research (CBPR) framework, which depends heavily upon community engagement and partnership throughout the entire research process, and Indigenous Food Sovereignty (IFS), a concept that represents Indigenous peoples' ability to control their food systems, including the production, distribution, and consumption of food. The Yup'ik word Yuuyaraq means 'the Yup'ik way of life' and it encompasses the Yup'ik worldview which is founded on traditional values of respect for humans, animals, and the environment in which they live, sharing of resources (including subsistence foods), sharing stories and knowledge, and an interpersonal relationship with nature as a source of wellness. The proposed intervention, Diet and Active Lifestyle- Yuuyaraq (DAiLY), is based on Yup'ik worldview principles.

DAiLY Intervention Components The intervention will be delivered through three complementary components, each supported and reinforced by community media, including social media (Facebook), texting and visual materials.

1. Home-Based Workshops (HBWs) will be delivered by trained members of the local community. The aim of the HBWs is to increase knowledge, skills and confidence related to to food (e.g., understanding nutrition labels, the benefits of traditional foods, supporting traditional subsistence and harvesting practices, making healthy market food choices, and healthy food preparation and serving methods), as well as participants' awareness of the importance of physical activity and maintaining a healthy weight. An emphasis is placed on understanding the benefits of consuming traditional subsistence foods, as well as heart-healthy foods from the local stores to complement the traditional diet.
2. Food store modifications will increase access to heart-healthy foods in local stores by working with store managers to stock and promote affordable healthy food options, which will in turn provide participants with the opportunity to implement what they have learned in the HBWs. Point of purchase promotions in stores, including educational displays, taste tests and cooking demonstrations, and temporary price reductions to build demand, will identify and promote these foods to community members.
3. Physical Activity (PA) opportunities will be increased, and will include community-based activities that have been identified by community members. These will emphasize traditional activities, such as Yuraq traditional Yup'ik Dance, Native sports events, and berry festivals. Fitbits will be given to participants and used as a motivational tool to encourage and allow participants to track their PA progress during and after the intervention.

Implementation and Assessment Community research associates (CRAs) will implement the DAiLY intervention after being trained by the study team, with follow-up booster trainings as needed. The intervention will be carried out in four communities, two of which will participate first (immediate intervention), allowing for comparison of outcomes among those who have and have not yet received the intervention. Once the follow-up data collection is complete, the second two communities (delayed intervention) will receive the intervention. Throughout all phases of the intervention, data will be collected about how well and to what extent the DAiLY intervention was implemented by the study team in each community.

The impact of the DAiLY intervention will be measured through changes in individual participants heart disease risk factors, as well as in the community food stores and in terms of access to increased PA opportunities at the community level. Participants will be asked to donate a fasting blood sample to measure the different factors that affect risk for heart disease, and study investigators (Boyer and Hopkins) will measure participants' weight, blood pressure and waist circumference. ActiGraph GT3X+, high-resolution triaxial accelerometers will be used to measure physical activity levels, in addition to completing a Yup'ik Wellness Questionnaire to assess participation in traditional and community activities and confidence to adopt healthy behaviors. In addition, a Yup'ik Food Frequency Questionnaire will be used to assess how participants report changes in dietary patterns and knowledge of healthy dietary behaviors. In community food stores, data will be collected on stocking and sales of promoted foods in store, as well as food store owners' and managers' expectations of sales of healthy food before and after the DAiLY intervention. We will also monitor changes in the availability, use (# people), PA quality and duration of community traditional PA opportunities. Physical activity opportunities in the community will be coordinated with the HBW modules and will include communityevents and subsistence activites. CRAs will receive $2000 per community to sponsor community-wide events. These activities will be initiated and promoted as part of the DAiLY including community campaigns to "park it and walk" to limit use of of snow machines and ATVs in the community, Fitbit step challenges, initiation of women's "walking groups" to gather their children at evening curfew, promotion of cultural events such as Yuraq traditional Yup'ik dance, holding berry festivals (including picking competitions) and supporting additional sports events (basketball, volleyball and Native games) in the school gyms. All of these community-level activities were suggested by our CPG.

Overall Project Aims Aim 1: Determine the effectiveness of the DAiLY intervention on HD risk by measuring: (1) change in a continuous metabolic syndrome (cMS) risk score (primary outcome) in Yup'ik adults; and (2) secondary outcomes including PA (using accelerometry), dietary change using objectively measured biomarkers, as well as dietary consumption, and change in psychosocial measures (i.e., knowledge, self-efficacy and intentions).

Aim 2: Assess implementation of the DAiLY intervention using a mixed methods process evaluation using a sequential explanatory design to determine: (1) reach, dose delivered, and fidelity; (2) barriers and facilitators to implementing program activities; and (3) participant satisfaction and engagement. Aim 3: Determine the impact of the DAiLY intervention on community-level outcomes including: (1) access to, and sales of, healthy foods in local stores; (2) access to community venues (e.g., school gyms and community halls for PA); and (3) frequency and level of engagement in subsistence activities and community-wide events.

Sharing Results and Dissemination of Program Materials A major objective of DAiLY is to share the results with the participating communities, as well as others who develop health promotion programs. The study team will continuously share the progress and results of the intervention with local community Tribal governments and healthcare leaders in order to ensure the communities that participated can determine next steps in their best interest. After completion of the trial, all intervention materials will be made available and freely downloadable from the study website.

ELIGIBILITY:
Inclusion Criteria:

* Participants Inclusion criteria: Self-identify as Yup'ik Alaska Native, Lives in a participating Yup'ik community, Does not plan to move out of the community throughout the intervention (24 months), 18 years of age or older.
* Communities Inclusion criteria: Willing to participate in the DAiLY intervention as evidenced by letters of support for the intervention study provided by community Tribal governments; Willing and ready to participate in the Community Based Participatory Research process (Community Planning Group, Home-based Workshops, Food Store Component, review of research outcomes) Food stores Inclusion Criteria: Located within the participating community, Store commonly used by community members, Does not anticipate closing permanently during the intervention period, Tribal Corporation stores (governed by Tribal Council) willing and able to facilitate all of the following intervention components at their food store: allow interactive sessions / taste tests in their food store, increase stocking of healthy foods and beverages, allow display of intervention shelf labels and other educational materials in their store (e.g., posters, flyers)

Exclusion Criteria:

* Participants Exclusion criteria: Currently pregnant (as dietary intake and PA recommendations differ during pregnancy), Anticipates moving out of the community in the next 24 months, Age is under 18 years of age, Participated in the pilot intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 368 (Estimated)
Dates: Start 2024-10-18 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-04-30 (Estimated)

PRIMARY OUTCOMES:
Continuous metabolic syndrome z score | From enrollment to the completion of post-intervention assessment (2 years)
  Determine the effectiveness of the DAiLY intervention on heart disease risk by measuring: (1) change in a continuous metabolic syndrome risk score (primary outcome) in Yup'ik adults at least 18 years old. The continuous metabolic syndrome score includes the weighted contributions of waist circumference, triglycerides, high density lipoprotein, glucose and blood pressure. The continuous metabolic syndrome score is a metabolic syndrome-severity Z score that adds predictive utility for future heart disease above and beyond the individual metabolic syndrome components.

SECONDARY OUTCOMES:
Dietary pattern change | From enrollment to the completion of post-intervention assessment (2 years)
  We will assess dietary consumption with a food frequency questionnaire validated for use in Yup'ik communities.
Moderate to Vigorous Physical Activity (MVPA) | From enrollment to the completion of post-intervention assessment, with a mid-point assessment (2 years)
  We will measure moderate to vigorous physical activity (MVPA) levels using accelerometry. Wrist-worn Actigraph GT3X+ monitors will be used. MVPA will be assessed using established wrist-worn accelerometry cutpoints and calculated as average minutes per day.
Knowledge | From enrollment to the completion of post-intervention assessment (2 years)
  The knowledge score assesses adult participants' knowledge of nutrition and physical activity (PA) behaviors emphasized in the intervention. Ten multiple choice questions cover topics such as dietary fiber, sugar, and nutrition label reading (alpha=0.63). An example is "Which kind of bread has the most fiber? a) Fry bread; b) White bread; c) 100% whole wheat bread; d) Don't know"
Self-efficacy | From enrollment to the completion of post-intervention assessment (2 years)
  The self-efficacy scale assesses the confidence that the respondent feels to carry out healthy physical activity and dietary behaviors. Eleven questions ask the respondent to categorize healthy behaviors as either "easy" or "difficult" within their lives (alpha=0.63). An example question is, "Would it be difficult or easy for you to choose water instead of regular soda?"
Intentions | From enrollment to the completion of post-intervention assessment (2 years)
  The healthy eating intentions score assesses a respondent's intention to perform healthy dietary or physical activity behaviors. Nine multiplechoice questions ask which of several food or activity options the respondent would select if they had to make a choice (alpha=0.60). An example question is "Next time you have free time at home, what will you do? a) Take a nap; b) Go for a walk or do housework; c) Watch TV or use the computer.
Nitrogen Isotope Ratio (NIR) | From enrollment to the completion of post-intervention assessment (2 years)
  The nitrogen isotope ratio(NIR) is assessed by measuring the ratio of 15N/14N in red blood cells.
Carbon Isotope Ratio (CIR) | From enrollment to the completion of post-intervention assessment (2 years)
  The carbon isotope ratio (CIR) is is assessed by measuring the ratio of 13C/12C.
Total Physical Activity | From enrollment to the completion of post-intervention assessment, with a mid-point assessment (2 years)
  We will measure total physical activity levels using accelerometry. Wrist-worn Actigraph GT3X+ monitors will be used.Total physical activity will be calculated using the average daily normal filtered vector magnitude counts using the ActiLife software.
Sedentary Time | From enrollment to the completion of post-intervention assessment, with a mid-point assessment (2 years)
  We will measure sedentary time using accelerometry. Wrist-worn Actigraph GT3X+ monitors will be used. Sedentary time will be assessed using established wrist-worn accelerometry cutpoints and calculated as average minutes per day.

OTHER OUTCOMES:
Reach | From beginning of intervention implementation to the completion of the intervention, about 2 years
  We will assess implementation of the DAiLY intervention by measuring reach of our trial. Reach refers to the number of individuals in the target audience participating in the intervention. Community Research Associates will document their work using structured Interventionist logs as they conduct each intervention component.
Community Impact | From beginning of intervention implementation to the completion of the intervention, about 2 years
  We will assess impact of the DAiLY intervention on community-level outcomes including: (1) access to, and sales of, healthy foods in local stores; and (2) access to community venues. We will modify a previously developed, successfully used, instrument for assessing the reported stocking and unit sales of promoted foods, outcome expectations of promoted food sales and effect of promotions on overall store sales and will be administered to store managers at two timepoints. A store food availability checklist form will be adapted for use in the Yupik community setting by including the specific foods and beverages that will be promoted for the DAiLY intervention. This instrument assesses availability of key promoted foods in food stores via a simple checklist and will be administered by the comm every two weeks in each of the community stores to allow for immediate midcourse correction where necessary. We will assess engagement in community events and school gym activities.
Dose Delivered | From beginning of intervention implementation to the completion of the intervention, about 2 years
  We will assess implementation of the DAiLY intervention by measuring the dose delivered of the trial. Dose delivered refers to the amount of time or the frequency that each activity is performed.
  Community Research Associates will document their work using structured Interventionist logs as they conduct each intervention component.
Fidelity | From beginning of intervention implementation to the completion of the intervention, about 2 years
  We will assess implementation of the DAiLY intervention by measuring fidelity. Fidelity refers to the engagement by the target audience in each of these activities.
  Community Research Associates will document their work using structured Interventionist logs as they conduct each intervention component.
Barriers to Intervention Implementation | From beginning of intervention implementation to the completion of the intervention, about 2 years
  We will assess implementation of the DAiLY intervention by determining barriers. Community Research Associates will document their work using structured Interventionist logs as they conduct each intervention component.
Facilitators for intervention implementation | From beginning of intervention implementation to the completion of the intervention, about 2 years
  We will assess implementation of the DAiLY intervention by identifying facilitators to implementation of program activities. Community Research Associates will document their work using structured Interventionist logs as they conduct each intervention component.
Participant Satisfaction | From beginning of intervention implementation to the completion of the intervention, about 2 years
  We will assess implementation of the DAiLY intervention through participant satisfaction. Community Research Associates will document their work using structured Interventionist logs as they conduct each intervention component. Focus groups will be conducted in each community after the homebased workshop series is complete to assess participant satisfaction.
Participant Engagement | From beginning of intervention implementation to the completion of the intervention, about 2 years
  We will assess implementation of the DAiLY intervention through participant engagement. Community Research Associates will document their work using structured Interventionist logs as they conduct each intervention component.

CONTACTS AND LOCATIONS:
Overall Officials: Bert B Boyer, PhD, Principal Investigator — Oregon Health and Science University
Locations (2):
- United States (2):
  - Yukon-Kuskokwim Health Corporation, Bethel, Alaska
  - Oregon Health and Science University, Portland, Oregon

IPD SHARING:
Plan to Share IPD: No
All individual participant data sharing is under the discretion of the Tribal Executive Board of the Yukon-Kuskokwim Health Corporation.

REFERENCES:
- [Background] O'Brien DM, Kristal AR, Nash SH, Hopkins SE, Luick BR, Stanhope KL, Havel PJ, Boyer BB. A stable isotope biomarker of marine food intake captures associations between n-3 fatty acid intake and chronic disease risk in a Yup'ik study population, and detects new associations with blood pressure and adiponectin. J Nutr. 2014 May;144(5):706-13. doi: 10.3945/jn.113.189381. Epub 2014 Mar 5. PMID 24598880
- [Background] Fienup-Riordan A. Eskimo Essays: Yup'ik Lives and How We See Them: Rutgers University Press; 1990.
- [Background] Ayunerak P, Alstrom D, Moses C, Charlie J Sr, Rasmus SM. Yup'ik culture and context in Southwest Alaska: community member perspectives of tradition, social change, and prevention. Am J Community Psychol. 2014 Sep;54(1-2):91-9. doi: 10.1007/s10464-014-9652-4. PMID 24771075
- [Background] Wolsko C, Lardon C, Hopkins S, Ruppert E. Conceptions of wellness among the Yup'ik of the Yukon-Kuskokwim Delta: the vitality of social and natural connection. Ethn Health. 2006 Nov;11(4):345-63. doi: 10.1080/13557850600824005. PMID 17060033
- [Background] Ray L, Burnett K, Cameron A, Joseph S, LeBlanc J, Parker B, Recollet A, Sergerie C. Examining Indigenous food sovereignty as a conceptual framework for health in two urban communities in Northern Ontario, Canada. Glob Health Promot. 2019 Apr;26(3_suppl):54-63. doi: 10.1177/1757975919831639. PMID 30964405
- [Background] Yu E, Malik VS, Hu FB. Cardiovascular Disease Prevention by Diet Modification: JACC Health Promotion Series. J Am Coll Cardiol. 2018 Aug 21;72(8):914-926. doi: 10.1016/j.jacc.2018.02.085. PMID 30115231
- [Background] Schwarz PEH, Timpel P, Harst L, Greaves CJ, Ali MK, Lambert J, Weber MB, Almedawar MM, Morawietz H. Reprint of: Blood Sugar Regulation for Cardiovascular Health Promotion and Disease Prevention: JACC Health Promotion Series. J Am Coll Cardiol. 2018 Dec 11;72(23 Pt B):3071-3086. doi: 10.1016/j.jacc.2018.10.026. PMID 30522637
- [Background] Micha R, Penalvo JL, Cudhea F, Imamura F, Rehm CD, Mozaffarian D. Association Between Dietary Factors and Mortality From Heart Disease, Stroke, and Type 2 Diabetes in the United States. JAMA. 2017 Mar 7;317(9):912-924. doi: 10.1001/jama.2017.0947. PMID 28267855
- [Background] Nash SH, Bersamin A, Kristal AR, Hopkins SE, Church RS, Pasker RL, Luick BR, Mohatt GV, Boyer BB, O'Brien DM. Stable nitrogen and carbon isotope ratios indicate traditional and market food intake in an indigenous circumpolar population. J Nutr. 2012 Jan;142(1):84-90. doi: 10.3945/jn.111.147595. Epub 2011 Dec 7. PMID 22157543
- [Background] Bersamin A, Luick BR, King IB, Stern JS, Zidenberg-Cherr S. Westernizing diets influence fat intake, red blood cell fatty acid composition, and health in remote Alaskan Native communities in the center for Alaska Native health study. J Am Diet Assoc. 2008 Feb;108(2):266-73. doi: 10.1016/j.jada.2007.10.046. PMID 18237575
- [Background] Boyer BB, Wiener HW, Hopkins SE, Purnell JQ, O'Brien DM, Aliwarga T, Pomeroy JJ, Aslan JE, Thummel KE, Tiwari HK. Obesity-Associated Dyslipidemia Is Moderated by Habitual Intake of Marine-Derived n-3 Polyunsaturated Fatty Acids in Yup'ik Alaska Native People: A Cross-Sectional Mediation-Moderation Analysis. J Nutr. 2023 Jan;153(1):279-292. doi: 10.1016/j.tjnut.2022.10.009. Epub 2022 Dec 21. PMID 36913463
- [Background] Alaska-Native-Epidemiology-Center. Alaska Native Mortality: 1980-2018. Anchorage: Alaska Native Tribal Health Consortium;2021.